CLINICAL TRIAL: NCT02968524
Title: Evaluation of Thermospot Accuracy in Nigerian Infants Exposed to Ambient Temperature and Validation of Maternal Readings and Responses
Acronym: Thermospot
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: HSR 16_4258
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: ThermoSpot Accuracy and Maternal Recognition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This project will focus on testing the accuracy of ThermoSpot -a low-cost, color-based, temperature indicator in estimating the body temperature of Nigerian babies exposed to ambient temperature conditions. The particpants will be recruited among babies receiving Filtered Sunlight Phototherapy (FSPT) at Bowen University Teaching Hospital, Ogbomoso and other babies in the nursery at Bowen University Teaching Hospital.

There will also be an educational session to teach health workers and mothers about the signs for hypothermia and hyperthermia on the indicator. Then, the investigators will collect observational cross-sectional data on random days to see how many of the trained health workers and mothers were able to accurately recognize and provide appropriate response to warning signs on the indicator.

DETAILED DESCRIPTION:
ThermoSpot is a liquid crystal display thermometer. It comes as a sticky disc (12mm in diameter) which can be applied to the skin over the liver, in the armpit, or over the neck blood vessels of an infant. ThermoSpot was designed as a non-invasive hypothermia indicator for infants. The device changes color when the baby's core body temperature changes, allowing it to be understood even by a non-literate parent. It has been tested and proven to accurately detect hypothermia in Malawi, Nepal and India. However, no large-scale studies have been performed on babies exposed to ambient temperatures for long periods such as those under FSPT.

The main objective of the project is to determine whether ThermoSpot can be used to detect hypothermia or hyperthermia in babies receiving FSPT instead of thermometers. The ability of a parent to respond in a timely manner to the temperature indicator will help provide critical information on technical, as well as educational components required for FSPT scale-up in Nigeria and other resource-limited countries with health worker shortage.

Specific objectives

1. Compare the performance of ThermoSpot in the detection of hypothermia or hyperthermia with the standard axillary thermometer measurement.
2. Determine if parents are able to correctly interpret the color indicators on ThermoSpot
3. Determine whether parents carry out the appropriate action based on the ThermoSpot indicator.

ELIGIBILITY:
Inclusion Criteria:

1. Babies under 4 weeks of age receiving FSPT (Infants ≥35wks gestation, or ≥2.2kg if gestational age is not available, and ≤14 days old at time of study enrollment), for whom parents or guardians have given consent to participate in the study.
2. Babies under 6 weeks of age in the nursery at Bowen University Teaching Hospital.
3. Parents or guardians of babies receiving FSPT who are interested in learning how to determine temperature using ThermoSpot and have given consent for their babies to participate in the study.

Exclusion Criteria:

1. Parental refusal
2. Infants already clinically dehydrated
3. Infants that are sunburned.

Max Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants 0-6 weeks who are either in the Filtered Sunlight Therapy Study or in the nursery at Bowen University Teaching Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Mother's Accuracy in using Thermospot | 1 year
  Will determine mother's ability to read the Thermospot and tell investigators the correct action needed if any

CONTACTS AND LOCATIONS:
Locations (1):
- Ogomo, Uganda

IPD SHARING:
Plan to Share IPD: No